CLINICAL TRIAL: NCT07249463
Title: A Randomized, Placebo-controlled, Participant- and Investigator-blinded Study to Assess the Efficacy and Safety and Tolerability of EDI048 in a Cryptosporidium Controlled Human Infection Model (CHIM) in Healthy Participants
Brief Title: Study Testing the Efficacy, Safety, and Tolerability of EDI048 in Cryptosporidium Infection Model in Healthy Adults
Acronym: CRYPTONITE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEDI048A12201
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cryptosporidiosis
Keywords: Cryptosporidiosis; Cryptosporidium; EDI048; ABO809; Controlled human infection model; CHIM
MeSH Terms: conditions — Cryptosporidiosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EDI048 (Experimental): Participants will receive ABO809 as a single oral dose. If participant is symptomatic, then he/she would be randomized to get EDI048 administered orally.
  Interventions: Biological: Cryptosporidium parvum oocysts (ABO809); Drug: EDI048
- Placebo (Placebo Comparator): Participants will receive ABO809 as a single oral dose. If participant is symptomatic, then he/she would be randomized to get placebo administered orally.
  Interventions: Biological: Cryptosporidium parvum oocysts (ABO809); Other: Placebo

INTERVENTIONS:
Biological: Cryptosporidium parvum oocysts (ABO809) — ABO809 oral suspension, single dose
Drug: EDI048 — EDI048 administered orally
  Arms: EDI048
Other: Placebo — Placebo administered orally
  Arms: Placebo

SUMMARY:
This study has the purpose to demonstrate prospect of benefit of EDI048 on clinical signs and symptoms of cryptosporidiosis to facilitate trial in target population, pediatric patients.

This study aims to investigate the efficacy of a new chemical entity, EDI048, in a controlled human infection model of cryptosporidiosis induced by administration of ABO809 in healthy adults, who become symptomatic with disease thereby demonstrating a prospect of benefit for use of EDI048 in children afflicted with cryptosporidiosis.

DETAILED DESCRIPTION:
This study is a Placebo-controlled, participant- and investigator-blinded multicenter trial in healthy adult volunteers who are administered Cryptosporidium parvum oocysts (ABO809) to develop diarrhea and symptoms consistent with cryptosporidiosis. After developing diarrhea, participants will be randomized 1:1 to treatment with EDI048 or placebo in parallel.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Ability to communicate well with the Investigator, and to understand and comply with the requirements of the study.
* Male and female participants must be between 18 to 50 years of age and in good health as determined by medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at Screening and Baseline.
* Demonstrate thorough understanding of cryptosporidiosis and measures to prevent secondary spread via education provided at screening.
* Must have a body mass index (BMI) within the range of 18-32 kg/m2. BMI = Body weight (kg) / [Height (m)]2
* Have not received ABO809 or EDI048 in prior clinical trials.

Exclusion Criteria:

* History of Cryptosporidium infection.
* Current (based on screening laboratory tests) or history of infectious diarrhea associated with international travel in the last 12 months or C. difficile infection within 6 months prior to Screening.
* Employment as a healthcare worker with direct patient care, in a daycare center (e.g., for children or the elderly), or direct food handler (individuals who work directly with food in commercial establishments).
* Participants who share a home with any of the following:
* a pregnant woman,
* a person <4 years old or >65 years old,
* a person who is infirmed,
* a person who is immunocompromised (for reasons including corticosteroid therapy, HIV infection, cancer chemotherapy, or other chronic debilitating disease).
* Residents of dormitories with shared bathrooms would also be excluded.
* Any significant medical history including, but not limited to, conditions of the cardiac, pulmonary, gastrointestinal, renal, endocrine, reproductive, immune or other systems.
* Use of investigational drugs within 5 half-lives of the drug or its major metabolites or 30 days of enrollment (Day 1), whichever is longer.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the trial; pregnant or nursing (lactating) women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-03-02 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
Average stool grade after the initiation of EDI048 or placebo treatment | Day 3, Day 4 and Day 5
  To determine the efficacy of EDI048 vs. placebo in healthy volunteers to reduce severity or resolve diarrhea.

SECONDARY OUTCOMES:
Maximum stool grade after the initiation of EDI048 or placebo treatment | Day 3, Day 4 and Day 5
  To determine the efficacy of EDI048 vs. placebo in healthy volunteers to reduce severity or resolve diarrhea.
Time to resolution of clinical diarrheal illness | up to Day 35
  To evaluate the efficacy of EDI048 vs. placebo based on signs and symptoms associated with clinical diarrheal characteristics.
Number of participants with associated gastrointestinal symptoms | up to Day 35
  To evaluate the efficacy of EDI048 vs. placebo based on signs and symptoms associated with clinical diarrheal characteristics.
Number of diarrhea episodes per participant | up to Day 35
  To evaluate the efficacy of EDI048 vs. placebo based on signs and symptoms associated with clinical diarrheal characteristics.
Overall diarrheal stool weight | up to Day 35
  To evaluate the efficacy of EDI048 vs. placebo based on signs and symptoms associated with clinical diarrheal characteristics.
Stool grade by stool grade category | up to Day 35
  To evaluate the efficacy of EDI048 vs. placebo based on signs and symptoms associated with clinical diarrheal characteristics.
Number of participants with fecal shedding of Cryptosporidium parvum oocysts | up to Day 35
  To evaluate the incidence of and time to resolution of Cryptosporidium infection in participants who received EDI048 vs. placebo.
Number of oocysts per gram per day (wet and dry weight) and the total number of oocyst per day measured by qPCR in fecal samples | up to Day 35
  To quantify fecal shedding of oocysts in participants who received EDI048 vs. placebo and to assess time to resolution of infection.
PK parameter: Cmax | up to Day 5
  To characterize PK of EDI048 and metabolite QPL621.
PK parameter: Tmax | up to Day 5
  To characterize PK of EDI048 and metabolite QPL621.
PK parameter: AUC0-t | up to Day 5
  To characterize PK of EDI048 and metabolite QPL621.
PK parameter: AUClast | up to Day 5
  To characterize PK of EDI048 and metabolite QPL621.
PK parameter: AUCinf | up to Day 5
  To characterize PK of EDI048 and metabolite QPL621.
PK parameter: T1/2 | up to Day 5
  To characterize PK of EDI048 and metabolite QPL621.
PK parameter: CI/F | up to Day 5
  To characterize PK of EDI048 and metabolite QPL621.
PK parameter: V/F | up to Day 5
  To characterize PK of EDI048 and metabolite QPL621.
Number of participants with adverse events of special interest (AESIs) | up to Day 35
  To assess the safety and tolerability of EDI048 vs. placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron Inc, Baltimore, Maryland, United States